CLINICAL TRIAL: NCT06149143
Title: Cardiac Performance System Data Collection Study - Minnesota
Status: Recruiting | Type: Observational
Sponsor: Sensydia Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CPS_MINNESOTA
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Function Monitoring: Subjects scheduled for cardiac catheterization will undergo measurement with the Cardiac Performance System non-invasive device for a brief period before the catheterization procedure.
  Interventions: Device: Cardiac Performance System (NSR)

INTERVENTIONS:
Device: Cardiac Performance System (NSR) — Participants will be asked to wear the Cardiac Performance System, a non-invasive sensor device on their upper abdomen. The Cardiac Performance System monitoring device will continuously monitor cardiac function.

SUMMARY:
Non-significant risk device study to conduct evaluation of the performance of new device for monitoring of cardiac function (based on previous iterations 510(k) 173156)

DETAILED DESCRIPTION:
Non-significant risk device study to conduct evaluation of the performance of new device for monitoring of cardiac function (based on previous iterations 510(k) 173156)

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* 22 years of age or older
* Referred for cardiac catheterization for reasons including heart failure, evaluation before transplant, pulmonary hypertension, shortness of breath, valvular disease, etc.

Exclusion Criteria:

* Previous Heart Transplant
* Presence of Left Ventricular Assist Device
* Presence of a Holter monitor or any other electrical leads on the chest at the time of sensor placement
* Surgical scars/wounds/bandages/ports at the site of sensor placement

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac catheterization procedure
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac Performance System electronic data for Cardiac Output | 10 minutes before cardiac catheterization procedure
  Cardiac function metric measurement including Cardiac Output to report in L/m.
Cardiac Performance System electronic data for Pulmonary Artery Pressure | 10 minutes before cardiac catheterization procedure
  Cardiac function metric measurement including Pulmonary Artery Pressure to report in mmHg.
Cardiac Performance System electronic data for Pulmonary Capillary Wedge Pressure | 10 minutes before cardiac catheterization procedure
  Cardiac function metric measurement including Pulmonary Capillary Wedge Pressure to report in mmHg.
Pulmonary Artery Catheter electronic data for Cardiac Output | 60 minutes during cardiac catheterization procedure
  Cardiac function metric measurement including Cardiac Output to report in L/m.
Pulmonary Artery Catheter electronic data for Pulmonary Artery Pressure | 60 minutes during cardiac catheterization procedure
  Cardiac function metric measurement including Pulmonary Artery Pressure to report in mmHg.
Pulmonary Artery Catheter electronic data for Pulmonary Capillary Wedge Pressure | 60 minutes during cardiac catheterization procedure
  Cardiac function metric measurement including Pulmonary Capillary Wedge Pressure to report in mmHg.
Echocardiography electronic data for Ejection Fraction | 15 minutes at a time prior to or after Pulmonary Artery Catheter procedure
  Cardiac function measurement including left ventricle ejection fraction to report in percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No